CLINICAL TRIAL: NCT00625859
Title: A Double-blind, Randomized, 6-sequence, 3-period, Crossover Drug Drug Interaction Study to Evaluate the Pharmacokinetics of Wellbutrin SR and GSK189075 When Co-administered or Administered Alone in Healthy Male Volunteers
Brief Title: A Study to Assess the Safety of Repeated Doses of GSK189075 and WELLBUTRIN SR in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: KGW111083
Record Dates: First submitted 2008-02-19; First posted 2008-02-28 (Estimated); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: pharmacodynamics; Healthy adult male volunteers,; pharmacokinetics,
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Bupropion

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Subjects receiving treatment sequence 1 (Experimental): Eligible subjects will receive treatment A in period 1, treatment B in period 2 and treatment C in period 3. A= Bupropion SR + GSK189075 placebo, B= Bupropion SR placebo + GSK189075 and C= Bupropion SR + GSK189075
  Interventions: Drug: GSK189075; Drug: Bupropion; Drug: Placebo
- Subjects receiving treatment sequence 2 (Experimental): Eligible subjects will receive treatment B in period 1, treatment C in period 2 and treatment A in period 3. A= Bupropion SR + GSK189075 placebo, B= Bupropion SR placebo + GSK189075 and C= Bupropion SR + GSK189075
  Interventions: Drug: GSK189075; Drug: Bupropion; Drug: Placebo
- Subjects receiving treatment sequence 3 (Experimental): Eligible subjects will receive treatment C in period 1, treatment A in period 2 and treatment B in period 3. A= Bupropion SR + GSK189075 placebo, B= Bupropion SR placebo + GSK189075 and C= Bupropion SR + GSK189075
  Interventions: Drug: GSK189075; Drug: Bupropion; Drug: Placebo
- Subjects receiving treatment sequence 4 (Experimental): Eligible subjects will receive treatment A in period 1, treatment C in period 2 and treatment B in period 3. A= Bupropion SR + GSK189075 placebo, B= Bupropion SR placebo + GSK189075 and C= Bupropion SR + GSK189075
  Interventions: Drug: GSK189075; Drug: Bupropion; Drug: Placebo
- Subjects receiving treatment sequence 5 (Experimental): Eligible subjects will receive treatment B in period 1, treatment A in period 2 and treatment C in period 3. A= Bupropion SR + GSK189075 placebo, B= Bupropion SR placebo + GSK189075 and C= Bupropion SR + GSK189075
  Interventions: Drug: GSK189075; Drug: Bupropion; Drug: Placebo
- Subjects receiving treatment sequence 6 (Experimental): Eligible subjects will receive treatment A in period 1, treatment C in period 2 and treatment B in period 3. A= Bupropion SR + GSK189075 placebo, B= Bupropion SR placebo + GSK189075 and C= Bupropion SR + GSK189075
  Interventions: Drug: GSK189075; Drug: Bupropion; Drug: Placebo

INTERVENTIONS:
Drug: GSK189075 — GSK189075 will be available as film-coated tablets with a dose of 250 milligrams.
Drug: Bupropion — Bupropion will be available as sustained release film-coated tablets with a dose of 150 milligrams administered orally.
Drug: Placebo — Placebo tablets will be given to subjects.

SUMMARY:
The purpose of this research study is to look at concentrations of GSK189075, WELLBUTRIN SR and active metabolic products in blood samples when doses of both drugs are taken by mouth. Doses are either taken alone or together. The results will help to determine if doses of GSK189075 and WELLBUTRIN SR can be safely taken together.

ELIGIBILITY:
INCLUSION CRITERIA:

* Healthy male subjects aged 18 to 55 years inclusive.
* Body Mass Index (BMI) is between 19-35kg/m2 (inclusive), with a minimum body weight of 45kg.
* Subject must read and write at a comprehension level that is sufficient to provide written informed consent, and be able to understand and comply with protocol requirements, instructions and protocol-stated restrictions.
* Subject has provided informed consent to participate in the study as indicated by providing a signed and dated written informed consent form prior to the initiation of any study procedures.

EXCLUSION CRITERIA:

* General

  * Presence of any clinically relevant abnormality identified on the screening medical assessment, laboratory examination or 12-lead ECG, or any other medical condition or circumstance making the volunteer unsuitable for participation in the study. These include any unstable medical disorder; disorders that would interfere with the action, absorption, distribution, metabolism, or excretion of bupropion or GSK189075; disorders which may pose a safety concern or interfere with the accurate assessment of safety or efficacy.
* Laboratory
* Clinically significant abnormalities at Screening including:

  * Systolic blood pressure outside the range of 90 - 140 mmHg, diastolic blood pressure outside the range of 50 - 90 mmHg, and pulse rate at rest > 100 and < 45 bpm.
  * Positive tests for hepatitis B surface antigen, hepatitis C antibodies, and HIV.
  * Positive cotinine, drug and/or alcohol test.
  * Significant ECG abnormalities are defined as follows:
* Parameter Range
* Heart Rate < 40 and >100 bpm
* PR Interval <120 and > 220 ms
* QRS duration < 70 and >120 ms
* QTC Interval (Bazett) > 450 ms

  * ALT, alkaline phosphatase, or total bilirubin ³ 1.5 times the upper limits of normal (Note: Subjects with an increased total bilirubin may enter the study only if direct bilirubin is within normal limits).
  * Fasting triglycerides >400 mg/dL (>11.3 mmol/L).
  * Clinically significant abnormalities of T3 and TSH.
  * Serum creatinine clearance <60ml/min (estimated from serum creatinine (SCr) and demographic data using the MDRD calculation):
* A validated web-based calculator is found at:
* http://nephron.com/cgi-bin/MDRDSIdefault.cgi
* To calculate estimated GFR (mL/min/1.73m2) manually:
* = 186 x (SCr in mg/dL)-1.154 x (age)-0.203 x (0.742 if female) x (1.210 if African-American)
* = exp(5.228-1.154 x ln (SCr)-0.203x ln(age)-(0.299 if female) + (0.192 if African American))

  * Any other clinically significant laboratory abnormality as determined by the Principal Investigator in consultation with the GSK Medical Monitor.
* Central Nervous System

  * Current diagnosis or a previous history of mania, psychosis, major depression, or other major psychiatric disorder.
  * Current or past history of seizure disorder or brain injury (traumatic or disease-related); or any condition which, in the opinion of the investigator, predisposes to seizure; those treated with other medications or treatment regimes that lower seizure threshold; those undergoing abrupt discontinuation of alcohol or sedatives (including benzodiazepines or benzodiazepine-like agents).
* Note: A single childhood febrile seizure is not exclusionary.

  * History or current diagnosis of anorexia nervosa or bulimia.
  * Subjects who, in the investigator's judgement, pose a homicidal or suicidal risk, have ever made a suicide attempt, or have ever been homicidal.
* Hepatic and Gastrointestinal systems

  * History of hepatic disease or known hepatic or biliary abnormalities, (with the exception of previously documented diagnosis of Gilbert's syndrome) and/or a history of biliary or gastrointestinal disorder, which might affect absorption, distribution, metabolism, or excretion of drugs (except appendectomy or cholecystectomy more than 12 weeks prior to the study).
* Endocrine system

  * Untreated or unstable thyroid disease. Subjects taking thyroid medications must be on a stable dosing regimen for at least 4 weeks prior to the first dose of study drug until completion of the Follow-up visit.
* Cardiac system

  * Subject has a history of clinically significant cardiac rhythm disorder or QTc interval ³450 milliseconds at Screening.
  * Subject has history of ischemic heart disease, including stable/unstable angina or acute myocardial infarction.
  * Uncontrolled hypertension with systolic blood pressure >140mm Hg and diastolic blood pressure >90mm Hg.

Drugs and Alcohol

* Subject has a history of alcohol abuse or an average weekly intake of greater than 21 units per week (one unit = 1 glass of wine = 1 measure of spirits = ½ pint of beer).
* Unwilling or unable to abstain from the use of illicit drugs and adhere to other protocol-stated restrictions while participating in the study.
* Use of tobacco in any form (smoking cigarettes, cigars, and/or pipes, or chewing tobacco-containing products), for 4 weeks prior to Screening until completion of the Follow-up visit.
* Unwilling or unable to abstain from the use of prescription or non-prescription drugs, vitamins, or dietary/herbal supplements within 1 week prior to the first dose of study drug until completion of the Follow-up visit.
* Subject is currently using medications that may alter gastric/small bowel motility, result in diarrhea, or bind concomitant medications. For example, but not limited to: erythromycin, antacids, prokinetic agents and cholestyramine.
* Subject has a history of drug or other allergy that, in the opinion of the Principal Investigator, contraindicates their participation in this study.

  • Concomitant medications usage that includes:
* Use of agents that are known to inhibit or induce cytochrome P450 enzymes within 14 days prior to the first dose of study medication , including grapefruit-containing products and St. John's Wort.
* Use of bupropion hydrochloride or GSK189075 within the last 6 months prior to Screening.
* Use of anti-depressant medication for clinically significant depression.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements within 7 days prior to the first dose in Treatment Period 1, unless in the opinion of the Investigator and Sponsor the medication will not interfere with the study procedures or compromise subject safety.

  * Note: Occasional use of acetaminophen and ibuprofen according to directions provided in the product label may be acceptable during the study, at the discretion of the Principal Investigator. Acetaminophen will be limited to doses up to 2 grams/day and ibuprofen at doses up to 1.2 grams/day.
  * Drug hypersensitivity
* History of hypersensitivity to WELLBUTRIN SR, ZYBAN, GSK189075 or any of their constituents or closely related compounds.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Other
* Past treatment with a new molecular entity (investigational drug) or any other trial during the previous 30 days, or 5 half-lives, whichever is longer. A new molecular entity is defined as any compound not in Phase 3. (The washout period of 30 days is counted from the last dose of study drug in the previous study until the first dose of study drug).
* Participation in the study would result in subject's donation of blood in excess of 500mL within a 56-day period.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2008-01-16 (Actual); Primary Completion 2008-04-10 (Actual); Study Completion 2008-04-10 (Actual)

PRIMARY OUTCOMES:
Blood samples and urine samples | on Day 14

SECONDARY OUTCOMES:
adverse events, heart rate & blood pressure: each visit ecg: screening, days -1, 1, 4, 7, 13, 14, followup lab tests: screening, days -1, 4, 7, 13, 14, followup | Up to Week 12
GSK189074 Cmax at steady-state when GSK189075 is administered alone and following co-administration with WELLBUTRIN SR. | Pre-dose, 0.25, 0.5, 1,2, 3, 4, 6, 8,10, 12, 16, 20 and 24hours
Bupropion and GSK189074 tmax at steady-state when GSK189075 is administered alone and following co-administration with WELLBUTRIN SR. | Pre-dose, 0.25, 0.5, 1,2, 3, 4, 6, 8,10, 12, 16, 20 and 24hours
Steady-state AUC(0-12), Cmax, and tmax of the bupropion metabolites (hydroxybupropion, threohydrobupropion and erythrohydrobupropion) when WELLBUTRIN SR is administered alone and with GSK189075. | Pre-dose, 0.25, 0.5, 1,2, 3, 4, 6, 8,10, 12, 16, 20 and 24hours
Steady-state AUC(0-12), Cmax, and tmax of GSK189075, and GSK279782 when GSK189075 is administered alone and with WELLBUTRIN SR. | Pre-dose, 0.25, 0.5, 1,2, 3, 4, 6, 8,10, 12, 16, 20 and 24hours
Safety and tolerability parameters, including adverse events (AEs), vital signs, ECGs and clinical laboratory assessments, including urine electrolytes (Na, Cl, K, Ca and Mg). | Pre-dose, 0.25, 0.5, 1,2, 3, 4, 6, 8,10, 12, 16, 20 and 24hours
Urine volume, urine glucose concentration, and urine creatinine concentration to determine fractional urine glucose excretion over a specified time interval (0-24h). | Up to Week 12
Hunger and craving will be assessed using two assessment tools: (1) a questionnaire to assess hunger and craving; and (2) a Visual Analogue Scale (VAS) to assess hunger. | Up to Week 12

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Buffalo, New York, United States

REFERENCES:
- See also: Results for study KGW111083 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/KGW111083?search=study&study_ids=KGW111083#rs